CLINICAL TRIAL: NCT02429427
Title: A Phase III Multicentre Double Blind Randomised Trial of Celecoxib Versus Placebo in Primary Breast Cancer Patients
Brief Title: European Celecoxib Trial in Primary Breast Cancer
Acronym: REACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C/20/01
Record Dates: First submitted 2015-04-15; First posted 2015-04-29 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
Keywords: Primary Breast Cancer; Celecoxib
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Celecoxib (Experimental): Patients in this arm will receive 400mg of celecoxib once daily. In addition, Hormone Receptor (+) patients will receive endocrine treatment according to local practice.
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Patients in this arm will receive 2 tablets once daily. In addition Hormone Receptor (+) patients will receive endocrine treatment according to local practice.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Celecoxib — Patients will receive 400mg of Celecoxib once daily for two years or until disease progression (if before the two years limit) or until development of unacceptable toxicities. In addition ER(+) patients will receive endocrine treatment according to local practice.
  Other Names: Celebrex, Onsenal, Celebra
  Arms: Celecoxib
Other: Placebo — Two capsules once daily with food
  Arms: Placebo

SUMMARY:
It has been found that the chemical changes that take place in a patient's body during the development of inflammation may provide an environment which stimulates cancer cells. One step in the development of inflammation is the production of certain chemical substances which are important in the formation and spread of tumours. These are called prostaglandins. Cyclo-oxygenase II (COX-2) is an enzyme (a substance that speeds up chemical changes in the body) involved in the production of these prostaglandins and although it is not usually present in most tissues it is made at the sites of inflammation. Celecoxib is a selective Non-Steroidal Anti Inflammatory Drug (NSAID) which works by blocking the action of the COX-2 enzyme, leading to a decrease in the production of prostaglandins and a reduction in inflammation.

The purpose of this study is therefore to find out if celecoxib can be used after breast cancer treatment (chemotherapy and/ or radiotherapy) to reduce inflammation and thus reduce the ability of new tumours to grow and survive.

2590 women with primary breast cancer will be recruited in this study from several locations in the United Kingdom and Germany. Eligible patients will be randomly allocated a treatment group, which can be celecoxib or placebo. Both treatments are taken orally (celecoxib 400mg daily, placebo 2 tablets daily) for a total of 2 years. In addition, hormone receptor positive patients will receive endocrine treatment as per local practice. Patients will prematurely discontinue treatment with celecoxib/placebo if disease progression is confirmed or if patients experience unacceptable toxicity.

Patients will be seen every 6 months for the first 3 years and then off treatment follow-up is carried out annually. Participating patients will also be given the option to take part in the pathology sub-study by donating a sample of the tumour tissue collected at the time of the primary surgery.

DETAILED DESCRIPTION:
It has long been recognised that there is an association between chronic immune activation and cancer but the mechanisms behind this observation are not fully understood. The inflammatory process may provide an environment for development of malignant disease, with mediators of inflammatory response such as the cyclo-oxygenases playing an important role and providing a target for therapeutic intervention.

Prostaglandins (PGs) are synthesised from phospholipids by the action of phospholipase A2 and cyclo-oxygenases. Cyclo-oxygenase (COX) -1 differs from COX-2 in that the latter is inducible and its expression is induced by a large range of oncogenes and growth factors. Celecoxib is a selective COX-2 inhibitor that does not cause the effects of COX-1 inhibition, namely gastrointestinal ulceration.

The key regulatory step in this process is the enzymatic conversion of fatty acids to PGG2 and PGH2 by COX. PGH2 is subsequently converted to one of several structurally related PGs including PGE2, PGD2, PGF2, and thromboxane A2 (TxA2), by the activity of specific PG synthases. PGs have important functions in every organ system and regulate a variety of physiological functions such as immunity, maintenance of vascular integrity and bone metabolism. COX-2 is not normally expressed in most tissues, but is induced by a wide spectrum of growth factors and pro-inflammatory cytokines in specific pathophysiological conditions. The expression of COX-2 is highly induced in cells transformed with the oncogene v-src or treated with phorbol esters.

Several studies have suggested an association between non-steroidal anti-inflammatory drug (NSAID) consumption and decreased breast cancer risk.

Elevated COX expression in breast cancer was suggested some time ago by the finding of elevated PG production in breast tumours.

There is pharmacological and genetic evidence to indicate that a significant component of the anticancer property of NSAIDs is due to their ability to inhibit the COX-2 enzyme.

This phase III randomised study assesses the impact on disease free survival and overall survival of the Cox-2 inhibitor Celecoxib as maintenance therapy following surgery and chemotherapy in the treatment of primary breast cancer.

2590 women with primary breast cancer will be recruited in this study from several locations in the United Kingdom and Germany.

Prior to randomization all patients should have completed at least 4 cycles of (neo) adjuvant chemotherapy. Patients who satisfy all the eligibility criteria for the study will be informed and consented to join the study. The Local Investigator will then contact the ICCG randomization centre to randomize the patient by fax or by telephone.

1. Assessments required pre-randomisation

   * Complete history and physical examination (within 4 weeks before randomisation)
   * Haematology (Hb, WBC or ANC, platelets) & Biochemistry [serum bilirubin, creatinine, alkaline phosphatase] (within 4 weeks before randomisation)
   * Mammogram, Chest X-ray, liver ultrasound, bone scan (at a maximum 00 months prior to diagnosis of breast cancer). In case of clinical symptoms metastatic disease has to be excluded before randomisation by the appropriate investigations
   * Collection of tissue blocks for the central tumour banks at Glasgow Royal Infirmary (for sites managed by ICCG) land Studienzentrale in Frankfurt (for sites managed by GBG)
2. Treatment

   Treatment must begin within 14 working days after randomisation and within 12 weeks of day 1 of the last cycle of adjuvant chemotherapy. Radiotherapy should be given according to local policy (concomitant trial treatment and radiotherapy is permitted). Patients will be randomised 2: 1 (in favour of celecoxib) to receive:

   Two Placebo capsules twice daily with food or Two Celecoxib 200mg capsules twice daily (800mg per day) with food The duration of celecoxib/placebo treatment is 2 years. In addition all postmenopausal ER + and/or PgR+ postmenopausal patients will receive exemestane (25mg daily) for 5 years. The start of the treatment will be at same time as starting celecoxib or placebo.
3. Routine Follow up Visits During the course of the trial all patients will be followed up every 3 months in the first year, every 6 months in !years 2 and 3 and annually from year 4 onwards.

   Follow up Assessments
   * Clinical examination and history
   * Haematology & biochemistry
   * Metastatic screen -additional tests/investigations (eg. Bone/liver scan etc) are at the investigators discretion if clinically indicated.
   * Serious Adverse Events
4. Follow up upon relapse Any relapse requires treatment to be stopped and patients should have the minimum tests carried out as described in section (c) above.

Relapse is categorized as ipsilateral breast or axillary nodal relapse [loco regional] distant relapse (including supraclavicular nodes) [distant] and contralateral breast disease (malignant) [2nd primary]. In the event of tumor recurrence the relevant recurrence form should be completed and the trials office notified within 4 weeks.

All patients will be followed up long term irrespective o whether they have been withdrawn from treatment prematurely.

ELIGIBILITY:
Inclusion Criteria:

1. Completely resected (greater or equal 1mm), histologically or cytologically proven unilateral breast cancer
2. Female greater or equal 18 years of age
3. If (neo) adjuvant chemotherapy received, patient must have received at least 4 cycles. Chemotherapy must be completed prior to study entry
4. Hormone Receptor negatives must have received prior chemotherapy
5. Study entry must be within any of the following timelines: 3 months of the end of definitive breast surgery OR between 3 weeks and 4 months after day 1 of the last cycle of adjuvant chemotherapy OR 6 weeks of the end of radiotherapy.
6. WHO performance status 0 or 1
7. Pre-treatment haematology and biochemistry values within acceptable local limits: Haemoglobin, white blood cell greater or equal to 3.0 x 109/l or absolute neutrophil count greater or equal to 1.51 x 109/l, Platelets greater or equal to 100 x 109/l, Serum bilirubin less than 1.5 x upper normal limit , Alkaline phosphatase less or equal to 1.5 x upper normal limit , Serum creatinine less than 1.5 x upper normal limit
8. Negative pregnancy test for patients with child-bearing potential
9. Normal baseline ECG and clinical cardiovascular assessment after completion of all (neo) adjuvant chemotherapy
10. No previous or current evidence for metastatic disease
11. Be accessible for and consent to long term follow-up
12. Written informed consent prior to commencement of specific protocol procedures must be obtained and documented according to the local regulatory requirements

Exclusion Criteria

1. Patients with node negative, T1, Grade 1 breast cancer
2. Unresectable, metastatic or bilateral breast cancer
3. Active or previous peptic ulceration or gastrointestinal bleeding in the last year
4. Active or previous history of inflammatory bowel disease
5. A past history of adverse reaction/hypersensitivity to NSAIDs, including celecoxib and salicylates, or sulphonamides
6. On current or planned chronic NSAIDs therapy (except low dose aspirin 100 mg four times per day or 325mg once daily).
7. Current or long-term use of oral corticosteroids
8. Known or suspected congestive heart failure (greater than New York Heart Association I) and/or coronary heart disease, previous history of myocardial infarction, uncontrolled arterial hypertension (ie BP greater than 160/90mmHg) under treatment with two anti-hypertensive drugs, rhythm abnormalities requiring permanent treatment.
9. Patients with diabetes controlled by diet and oral medication are eligible for the study however patients with insulin dependent diabetes are excluded
10. Past history of stroke/Transient ischaemic attack, symptomatic peripheral vascular disease or carotid disease
11. Previously entered into an adjuvant chemotherapy trial for which approval for entry into REACT has not been granted
12. ER receptor status unknown, Human epidermal growth factor receptor 2 or FISH positive, or Human epidermal growth factor receptor 2 status unknown

14. Hormone Receptor negative and not received (neo)adjuvant chemotherapy 15. Use of hormone replacement therapy within the last 6 weeks 16. Pregnant or lactating women or women of childbearing potential unwilling/unable to use non-hormonal contraception 17. No previous or concomitant malignancies except adequately treated squamous cell / basal cell carcinoma of the skin, in situ carcinoma of the cervix or ductal carcinoma in situ/lobular carcinoma in situ of the breast, unless there has been a disease-free interval of 10 years or more 18. Psychiatric or addictive disorders which could preclude obtaining informed consent 19. Clinical evidence of severe osteoporosis and/or history of osteoporotic fracture

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2639 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Coombes, MD, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coombes RC, Tovey H, Kilburn L, Mansi J, Palmieri C, Bartlett J, Hicks J, Makris A, Evans A, Loibl S, Denkert C, Murray E, Grieve R, Coleman R, Borley A, Schmidt M, Rautenberg B, Kunze CA, Rhein U, Mehta K, Mousa K, Dibble T, Lu XL, von Minckwitz G, Bliss JM; Randomized European Celecoxib Trial (REACT) Trial Management Group and Investigators. Effect of Celecoxib vs Placebo as Adjuvant Therapy on Disease-Free Survival Among Patients With Breast Cancer: The REACT Randomized Clinical Trial. JAMA Oncol. 2021 Sep 1;7(9):1291-1301. doi: 10.1001/jamaoncol.2021.2193. PMID 34264305
- See also: REACT Trial Information linked to the sponsor webpage — http://www1.imperial.ac.uk/cancer/iccg/breast/react/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Celecoxib | Placebo
Started | 1763 | 876
Completed | 1392 | 697
Not Completed | 371 | 179
Not completed — Adverse Event | 220 | 92
Not completed — Protocol Violation | 10 | 6
Not completed — Lost to Follow-up | 15 | 6
Not completed — Withdrawal by Subject | 64 | 34
Not completed — Other | 62 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Placebo | Total
Number analyzed (Participants) | 1763 | 876 | 2639
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55.2 [48.7 to 62.6] | 55.3 [48.6 to 63.0] | 55.2 [48.6 to 62.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1763 | 876 | 2639
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 1689 | 848 | 2537
  Ethnicity: Asian | 29 | 8 | 37
  Ethnicity: Other | 21 | 10 | 31
  Ethnicity: Black Caribbean | 13 | 4 | 17
  Ethnicity: Black African | 8 | 4 | 12
  Ethnicity: Black Other | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS) Benefit of Two Years Adjuvant Therapy With the COX-2 Inhibitor Celecoxib Compared With Placebo in Primary Breast Cancer Patients.
Description: From time of randomisation to the date of first event; with events contributing to the analysis defined as loco-regional and distant breast cancer recurrence, new primary breast cancer (ipsilateral or contralateral) and death without disease relapse (intercurrent death)
Time Frame: Patients will be followed up to 10 years. DFS will be calculated from date of randomization until the date of first documented DFS event, this will be assessed at 2 and 5 years
Population: Intention To Treat: This population includes all patients entered into the study in the treatment group they were allocated to regardless of whether they do not start treatment, take the wrong treatment or deviate in any way from the protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 1763 | 876
Percentage of participants
  2 Year DFS rate | 91 [90 to 93] | 90 [87 to 92]
  5 Year DFS rate | 84 [82 to 86] | 83 [81 to 86]
Statistical Analysis 1: Comparison: Celecoxib vs Placebo; Test type: Superiority; p = 0.751, Log Rank; Analysis stratified by oestrogen receptor status and country; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.80 to 1.17] — Analysis stratified by oestrogen receptor status and country

2. Secondary Outcome: Overall Survival
Description: First local recurrence and first distant recurrence will be recorded on separate parts of the CRF. In the event of local progression, all patients must be followed up for distant recurrence, second malignancy and survival. Similarly in the case of second malignancy, the appropriate CRF should be completed and patients should REACT Protocol, Version 39, dated 01.11.2016 Page 34 of 48 continue to be followed for disease progression and where possible the relation of any subsequent disease progression and/or death due to the primary or second cancer should be established.
Time Frame: Date of randomisation until the date of death from any cause or censored at the date the patient was last seen alive, this will be assessed at 2 and 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 1763 | 876
Percentage of participants
  2 Year | 97 [96 to 97] | 96 [95 to 97]
  5 Year | 90 [89 to 92] | 91 [88 to 92]
Statistical Analysis 1: Comparison: Celecoxib vs Placebo; Test type: Superiority; p = 0.781, Log Rank; Analysis is stratified for oestrogen receptor status and country; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.76 to 1.22] — Analysis is stratified for oestrogen receptor status and country

3. Secondary Outcome: Number of Participants With Incidence of Second Primary Breast Cancers
Description: Any malignant contralateral breast disease will be included and recorded as a second primary
Time Frame: From randomisation until a second primary breast cancer is diagnosed. Patients will be followed up to 10 years.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 1763 | 876
Participants | 19 | 12

4. Secondary Outcome: Cardiovascular Mortality
Description: Number of deaths recorded as having cardiovascular involvement are reported by treatment group.
Time Frame: Patients are followed up to 10 years, any deaths within this timeframe with cardiovascular involvement reported are included in the analysis.
Population: Safety population: This population includes all patients who start treatment, patients will be analysed by the treatment they received regardless of the group they were allocated to.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 1755 | 868
Participants | 6 | 5

ADVERSE EVENTS:
Time Frame: From the time of randomisation until 30 days after the discontinuation of celecoxib/placebo (i.e. 2 years or sooner if patient discontinued early).
Description: Only adverse events classed as grade 2 or above were collected. Adverse Events and SAEs were assessed in the Safety Population and All-Cause Mortality was assessed for all enrolled participants
Arm/Group | Celecoxib | Placebo
All-Cause Mortality (participants affected / at risk) | 203/1763 | 104/876
Serious Adverse Events (participants affected / at risk) | 148/1755 | 64/868
Other Adverse Events (participants affected / at risk) | 298/1755 | 151/868
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib (N=1755) | Placebo (N=868)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute cardiac event (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 7 (7) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 6 (6) | 2 (2)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 1 (1)
Fibrosis (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Perforated ulcer (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Suprapubic pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 3 (3) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 7 (9) | 2 (2)
Infection (Infections and infestations) | 6 (9) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Mastitis (Infections and infestations) | 3 (3) | 2 (2)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Uterine infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 2 (2) | 0 (0)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Clavicle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Foot fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Humerus fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lower limb fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Radius fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tibia fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 3 (3)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (4) | 4 (4)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Psychiatric symptom (Psychiatric disorders) | 3 (3) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Adnexal torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast necrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erysipelas (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling of eyelid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0)
Breast reconstruction (Surgical and medical procedures) | 3 (3) | 2 (4)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Oophorectomy bilateral (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Epistaxis (Vascular disorders) | 1 (1) | 0 (0)
Haematemesis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Myocardial infarction (Vascular disorders) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=1755) | Placebo (N=868)
Arthralgia (Musculoskeletal and connective tissue disorders) | 128 | 85
Hot flush (Reproductive system and breast disorders) | 106 | 54
Hypertension (Vascular disorders) | 178 | 72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT02429427/Prot_000.pdf
  • Statistical Analysis Plan (2014-06-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT02429427/SAP_001.pdf